CLINICAL TRIAL: NCT05366127
Title: Validation of a Simplified Severity Score (Investigator Global Assessment: IGA) in Bullous Pemphigoid
Acronym: IGA score
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0017/OB
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with bullous pemphigoid: IGA score and BPDAI score will be assessed to patient with bullous pemphigoid
  Interventions: Other: IGA score; Other: BULLOUS PEMPHIGOID DISEASE AREA INDEX (BPDAI)

INTERVENTIONS:
Other: IGA score — IGA score will be assessed by 2 blinded investigators
Other: BULLOUS PEMPHIGOID DISEASE AREA INDEX (BPDAI) — BPDAI will be assessed by 2 by 2 blinded investigators

SUMMARY:
The aim of the study is to validate a global and simple score : IGA (Investigator Global Assessment) score for the evaluation of the extent and severity of the disease in patients with bullous pemphigoid

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients aged ≥ 18 years
* Newly diagnosed or relapsing BP
* Clinical features suggestive of classic BP AND suggestive histological features AND deposition of IgG and/ or C3 deposits on the dermal epiderma junction, AND detection of circulating anti-epidermal antibodies labelling the epidermal side of salt-split skin
* Patient having read and understood the information letter and not opposed to participation
* Must be willing and able to adhere to all specified requirements, including but not limited to adherence to the follow-up visits

Exclusion Criteria:

* Predominant or exclusive mucosal involvement leading to suspect the diagnosis of mucous membrane pemphigoid
* Pemphigoid gestationis
* Linear IgA dermatosis (predominant or exclusive IgA deposits on the DEJ)
* Skin lesions suggesting the diagnosis of epidermolysis bullosa acquisita (skin fragility, atrophy, milia)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with bullous pemphigoid
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of IGA Score between baseline and 6-month follow-up visit | 6 months
  IGA score : 0 to 4
BPDAI Score between baseline and 6-month follow-up visit | 6 months
  BPDAI : 0 to 120

SECONDARY OUTCOMES:
Evolution of IGA Score between baseline and 3-month follow-up visit | 3 months
  IGA score : 0 to 4
Evolution of IGA Score between baseline and 2-month follow-up visit | 2 months
  IGA score : 0 to 4
Evolution of IGA Score between baseline and 1-month follow-up visit | 1 month
  IGA score : 0 to 4
Evolution of IGA Score between baseline and 3-weeks follow-up visit | 3 weeks
  IGA score : 0 to 4
Evolution of IGA Score between baseline and 2-weeks follow-up visit | 2 weeks
  IGA score : 0 to 4
Evolution of IGA Score between baseline and 1-week follow-up visit | 1 week
  IGA score : 0 to 4
Evolution of BPDAI Score between baseline and 3-month follow-up visit | 3 months
  BPDAI : 0 to 120
Evolution of BPDAI Score between baseline and 2-month follow-up visit | 2 months
  BPDAI : 0 to 120
Evolution of BPDAI Score between baseline and 1-month follow-up visit | 1 month
  BPDAI : 0 to 120
Evolution of BPDAI Score between baseline and 3 weeks follow-up visit | 3 weeks
  BPDAI : 0 to 120
Evolution of BPDAI Score between baseline and 2 weeks follow-up visit | 2 weeks
  BPDAI : 0 to 120
Evolution of BPDAI Score between baseline and 1 week follow-up visit | 1 week
  BPDAI : 0 to 120

CONTACTS AND LOCATIONS:
Overall Officials: Pascal JOLY, Principal Investigator — University Hospital, Rouen
Locations (11):
- France (11):
  - Bordeaux University Hospital, Bordeaux
  - Dijon University Hospital, Dijon
  - Lille University Hospital, Lille
  - Lyon University Hospital, Lyon
  - Montpellier University Hospital, Montpellier
  - Nantes University Hospital, Nantes
  - Avicennes Hospital, Paris
  - Bichat Hospital, Paris
  - Henri Mondor Hospital, Paris
  - Saint-Louis Hospital, Paris
  - Reims University Hospital, Reims

IPD SHARING:
Plan to Share IPD: No